CLINICAL TRIAL: NCT07315997
Title: The Coronary Artery Calcium and Troponins in Rheumatoid Arthritis (CAT-RA) Study
Acronym: CAT-RA
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Katherine P Liao, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2024P001981
Record Dates: First submitted 2025-12-31; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis (RA; Atherosclerotic Cardiovascular Disease (ASCVD)
Keywords: CAT-RA
MeSH Terms: conditions — Arthritis, Rheumatoid; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: high sensitivity cardiac troponin — Blood measurement of high sensitivity cardiac troponin

SUMMARY:
Individuals with rheumatoid arthritis (RA) have up to 2x the risk of having a heart attack compared to someone without RA. The goal of this study is to identify biomarkers that can help us do a better job of identifying individuals at risk before they develop symptoms of heart disease and start preventative treatment earlier.

DETAILED DESCRIPTION:
The objective of this study is to test the utility of high sensitivity cardiac troponin (hs-cTn) and coronary artery calcium (CAC) in risk stratifying patients with rheumatoid arthritis (RA) who may benefit from lipid lowering therapy. The population of interest are individuals who would not otherwise be recommended for therapy based on general population risk calculators for heart disease risk.

ELIGIBILITY:
Inclusion Criteria:

* RA diagnosed by a rheumatologist
* Age 40- 79
* ≥1 ASCVD risk factor including prediabetes, hypertension, BMI >30, current or history of cigarette smoking

Exclusion Criteria:

* Patients on a statin or with a contraindication to statin, on a cholesterol absorption inhibitor, or on a PCSK9 inhibitor
* Patients with diabetes mellitus
* Pregnancy

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with rheumatoid arthritis, age 40- 79 years, with one cardiovascular risk factor and not on a statin or has a contraindication to statin therapy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2028-03-04 (Estimated); Study Completion 2028-03-04 (Estimated)

PRIMARY OUTCOMES:
coronary artery calcium score | Cross-sectional, at baseline
  Quantified coronary artery calcium score

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Pending IRB approval.